CLINICAL TRIAL: NCT00271596
Title: A Randomized, Placebo-Controlled Pilot Study in Huntington's Disease (CIT-HD)
Brief Title: Citalopram to Enhance Cognition in HD
Acronym: CIT-HD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Cure Huntington's Disease Initiative (CHDI) (Unknown); University of Rochester (Other); Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jess G. Fiedorowicz, Assistant Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200509746; 5K23NS055733 (NIH); A-2063 (Other: CHDI Foundation)
Record Dates: First submitted 2005-12-30; First posted 2006-01-02 (Estimated); Results first posted 2013-03-13 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-02

CONDITIONS: Huntington Disease; Chorea; Executive Dysfunction
Keywords: Huntington Disease; Citalopram; Celexa; Chorea; Focus; ADD; ADHD; HD; SSRI
MeSH Terms: conditions — Huntington Disease; Chorea; Attention Deficit Disorder with Hyperactivity | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Citalopram (Experimental): 20mg daily citalopram
  Interventions: Drug: 20mg daily citalopram
- Placebo (Placebo Comparator): Matching daily placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 20mg daily citalopram — a selective serotonin reuptake inhibitor (SSRI) treatment administered over 16 weeks
  Other Names: Celexa
  Arms: Citalopram
Drug: Placebo — a daily matching placebo administered over 16 weeks
  Other Names: Matching daily placebo
  Arms: Placebo

SUMMARY:
This research plan proposes to conduct a double-blind, placebo-controlled pilot clinical trial in 36 adults with mild Huntington's disease (HD) to address the following research aims:

1. To determine the effect of citalopram compared to placebo in patients with early HD on executive function and other outcome variables including functional measures (health-related quality of life, work productivity, and self-reported attention), motor performance, and psychiatric status,
2. To study the relationship between executive function and functional status in patients with early HD after selective serotonin reuptake inhibitor (SSRI) treatment, and
3. To examine the effect of citalopram treatment on volumetric and metabolic (i.e, N-acetyl-aspartate concentration) measures in the neostriatum among patients with recently diagnosed Huntington's disease.

DETAILED DESCRIPTION:
Specific Aims:

1. To examine the effects of sixteen weeks of treatment with the selective serotonin reuptake inhibitor (SSRI) citalopram compared to placebo on executive function in patients with early Huntington's disease (HD).
2. To study the relationship between executive function and functional status in patients with early HD after SSRI treatment.
3. To determine the effect of sixteen weeks of citalopram compared to placebo on other outcome variables including functional measures (health-related quality of life, work productivity, and self-reported attention), motor performance, and psychiatric status.
4. To examine the effect of citalopram treatment on volumetric and metabolic (i.e, N-Acetyl-Aspartate concentration) measures in the neostriatum among patients with recently diagnosed Huntington's Disease.

Main Hypotheses:

1. At the end of the treatment protocol, patients receiving citalopram as compared with placebo will show a significantly greater improvement on tests of executive function.
2. Performance on measures of executive function will be significantly associated with measures of functional status.
3. At the end of the treatment protocol, patients receiving citalopram as compared with placebo will show a significantly greater improvement in functional status and psychiatric ratings; motor score is not expected to change as a result of citalopram therapy.
4. Using structural MRI and occipital proton magnetic resonance spectroscopy (1H-MRS), after treatment, patients with recently diagnosed Huntington's Disease will show greater changes from baseline on volumetric and metabolic (i.e., N-Acetyl-Aspartate concentration) neuroimaging measures in the neostriatum than those on placebo.

ELIGIBILITY:
Inclusion Criteria:

* Gene positive HD test (or, if untested, an HD diagnosis) with some abnormal motor signs (i.e., diagnostic confidence level of greater than or equal to 1 as measured by the UHDRS).
* Aged between 18 and 75
* Ability to provide written informed consent
* Mild stage HD (Shoulson and Fahn Scale Stage 1 or 2)
* Mild executive dysfunction: Participants must have complaints of poor cognition, mild functional decline, or demonstrate objective evidence of decline from their premorbid level
* Participants are able to complete all study assessments

Exclusion Criteria:

* Age under 18 or greater than 75
* Current major depression deemed significant by the investigator at the screening visit or current suicidal ideation.
* Any unstable or severe psychiatric disease including diagnoses of schizophrenia, bipolar affective disorder, dementia, delirium, severe anxiety and/or substance abuse/dependence.
* Current use of an SSRI or other treatment for depression (e.g., use of an MAOI) or treatment with an SSRI within the past 14 days.
* Current use of St. John's wort within the past 14 days.
* To ensure performance on cognitive measures are not affected by specific concomitant medications, participants taking methylphenidate, amphetamine/dextroamphetamine, atomoxetine, an acetyl cholinesterase inhibitor, an atypical antipsychotic, kava kava, Ginkgo Biloba, or an anxiolytic drug may be excluded unless their dose and dosing frequency have remained stable for 30 days prior to receiving study drug. Continued participation also requires the dose and dosing frequency remain stable throughout the study.
* Patients who are pregnant, nursing, or planning to become pregnant during the study.
* Patients who are unable to participate in the study assessments (cognitive, functional, psychiatric and motor scales) due to cognitive, motor, or sensory impairments (i.e., significant vision or hearing deficits).
* Other serious medical conditions such as cardiovascular or cerebrovascular disease; head injury deemed clinically significant by the PI; neurological disorder or insult other than HD.
* Learning disability or other medical condition that is likely to affect cognitive function; history of symptoms indicative of attention deficit hyperactivity disorder (ADHD) in childhood; or a diagnosis of ADHD.

It is important to note that participants who are unable to receive an MRI scan may still participate in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2005-11; Primary Completion 2011-04 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leigh J Beglinger, Ph.D., Principal Investigator — The University of Iowa Psychiatry Department; Jess G Fiedorowicz, M.D., Ph.D., Principal Investigator — University of Iowa Psychiatry Department; Kevin Biglan, M.D., M.P.H., Principal Investigator — University of Rochester; John Caviness, M.D., Principal Investigator — Mayo Clinic; Ricardo Jorge, M.D., Principal Investigator — University of Iowa Psychiatry Department
Locations (3):
- United States (3):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - The University of Iowa, Iowa City, Iowa
  - University of Rochester, Rochester, New York

REFERENCES:
- [Background] Aylward EH, Anderson NB, Bylsma FW, Wagster MV, Barta PE, Sherr M, Feeney J, Davis A, Rosenblatt A, Pearlson GD, Ross CA. Frontal lobe volume in patients with Huntington's disease. Neurology. 1998 Jan;50(1):252-8. doi: 10.1212/wnl.50.1.252. PMID 9443488
- [Background] Bauer A, Zilles K, Matusch A, Holzmann C, Riess O, von Horsten S. Regional and subtype selective changes of neurotransmitter receptor density in a rat transgenic for the Huntington's disease mutation. J Neurochem. 2005 Aug;94(3):639-50. doi: 10.1111/j.1471-4159.2005.03169.x. PMID 16033418
- [Background] Bonelli RM, Wenning GK, Kapfhammer HP. Huntington's disease: present treatments and future therapeutic modalities. Int Clin Psychopharmacol. 2004 Mar;19(2):51-62. doi: 10.1097/00004850-200403000-00001. PMID 15076012
- [Background] Como PG, Rubin AJ, O'Brien CF, Lawler K, Hickey C, Rubin AE, Henderson R, McDermott MP, McDermott M, Steinberg K, Shoulson I. A controlled trial of fluoxetine in nondepressed patients with Huntington's disease. Mov Disord. 1997 May;12(3):397-401. doi: 10.1002/mds.870120319. PMID 9159735
- [Background] Duan W, Guo Z, Jiang H, Ladenheim B, Xu X, Cadet JL, Mattson MP. Paroxetine retards disease onset and progression in Huntingtin mutant mice. Ann Neurol. 2004 Apr;55(4):590-4. doi: 10.1002/ana.20075. PMID 15048901
- [Background] Fennema-Notestine C, Archibald SL, Jacobson MW, Corey-Bloom J, Paulsen JS, Peavy GM, Gamst AC, Hamilton JM, Salmon DP, Jernigan TL. In vivo evidence of cerebellar atrophy and cerebral white matter loss in Huntington disease. Neurology. 2004 Sep 28;63(6):989-95. doi: 10.1212/01.wnl.0000138434.68093.67. PMID 15452288
- [Background] Kish SJ, Shannak K, Hornykiewicz O. Elevated serotonin and reduced dopamine in subregionally divided Huntington's disease striatum. Ann Neurol. 1987 Sep;22(3):386-9. doi: 10.1002/ana.410220318. PMID 2445259
- [Background] Menza M, Marin H, Kaufman K, Mark M, Lauritano M. Citalopram treatment of depression in Parkinson's disease: the impact on anxiety, disability, and cognition. J Neuropsychiatry Clin Neurosci. 2004 Summer;16(3):315-9. doi: 10.1176/jnp.16.3.315. PMID 15377738
- [Background] Murman DL, Giordani B, Mellow AM, Johanns JR, Little RJ, Hariharan M, Foster NL. Cognitive, behavioral, and motor effects of the NMDA antagonist ketamine in Huntington's disease. Neurology. 1997 Jul;49(1):153-61. doi: 10.1212/wnl.49.1.153. PMID 9222184
- [Background] Naarding P, Kremer HP, Zitman FG. Huntington's disease: a review of the literature on prevalence and treatment of neuropsychiatric phenomena. Eur Psychiatry. 2001 Dec;16(8):439-45. doi: 10.1016/s0924-9338(01)00604-6. PMID 11777733
- [Background] Patel SV, Tariot PN, Asnis J. L-Deprenyl augmentation of fluoxetine in a patient with Huntington's disease. Ann Clin Psychiatry. 1996 Mar;8(1):23-6. doi: 10.3109/10401239609149087. PMID 8743645
- [Background] Ranen NG, Lipsey JR, Treisman G, Ross CA. Sertraline in the treatment of severe aggressiveness in Huntington's disease. J Neuropsychiatry Clin Neurosci. 1996 Summer;8(3):338-40. doi: 10.1176/jnp.8.3.338. PMID 8854307
- [Background] Reynolds GP, Dalton CF, Tillery CL, Mangiarini L, Davies SW, Bates GP. Brain neurotransmitter deficits in mice transgenic for the Huntington's disease mutation. J Neurochem. 1999 Apr;72(4):1773-6. doi: 10.1046/j.1471-4159.1999.721773.x. PMID 10098889
- [Background] Reynolds GP, Pearson SJ. Decreased glutamic acid and increased 5-hydroxytryptamine in Huntington's disease brain. Neurosci Lett. 1987 Jul 22;78(2):233-8. doi: 10.1016/0304-3940(87)90639-2. PMID 2442679
- [Background] Rosas HD, Koroshetz WJ, Chen YI, Skeuse C, Vangel M, Cudkowicz ME, Caplan K, Marek K, Seidman LJ, Makris N, Jenkins BG, Goldstein JM. Evidence for more widespread cerebral pathology in early HD: an MRI-based morphometric analysis. Neurology. 2003 May 27;60(10):1615-20. doi: 10.1212/01.wnl.0000065888.88988.6e. PMID 12771251
- [Background] Shoulson I, Goldblatt D, Charlton M, Joynt RJ. Huntington's disease: treatment with muscimol, a GABA-mimetic drug. Ann Neurol. 1978 Sep;4(3):279-84. doi: 10.1002/ana.410040316. PMID 152602
- [Background] Yohrling IV GJ, Jiang GC, DeJohn MM, Robertson DJ, Vrana KE, Cha JH. Inhibition of tryptophan hydroxylase activity and decreased 5-HT1A receptor binding in a mouse model of Huntington's disease. J Neurochem. 2002 Sep;82(6):1416-23. doi: 10.1046/j.1471-4159.2002.01084.x. PMID 12354289
- [Derived] Beglinger LJ, Adams WH, Fiedorowicz JG, Duff K, Langbehn D, Biglan K, Caviness J, Olson B, Paulsen JS. Practice Effects and Stability of Neuropsychological and UHDRS Tests Over Short Retest Intervals in Huntington Disease. J Huntingtons Dis. 2015;4(3):251-60. doi: 10.3233/JHD-150159. PMID 26444022
- [Derived] Beglinger LJ, Adams WH, Langbehn D, Fiedorowicz JG, Caviness J, Biglan K, Olson B, Paulsen JS. Does interval between screening and baseline matter in HD cognitive clinical trials? J Huntingtons Dis. 2014;3(2):139-44. doi: 10.3233/JHD-140100. PMID 25062857
- [Derived] Beglinger LJ, Adams WH, Langbehn D, Fiedorowicz JG, Jorge R, Biglan K, Caviness J, Olson B, Robinson RG, Kieburtz K, Paulsen JS. Results of the citalopram to enhance cognition in Huntington disease trial. Mov Disord. 2014 Mar;29(3):401-5. doi: 10.1002/mds.25750. Epub 2013 Dec 27. PMID 24375941
- See also: The University of Iowa's Huntington's Disease Center of Excellence — http://www.uihealthcare.com/depts/huntingtonsdisease/index.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-six individuals were screened and 33 participants were randomized between May 2007 and April 2011 Participants were recruited using advertisements, by speaking at HD events, through local clinics and through two HD registries: The University of Iowa HD registry and the National HD Research Roster (Indiana).
Pre-assignment Details: Following the baseline visit, participants completed a study visit (i.e., Visit 01) after 2 weeks in order to wash-out practice effects on primary outcome measures. To further control for practice effects, participants received placebo for 14 days prior to randomization (i.e., using a placebo run-in design).
Period: Overall Study
Arm/Group | Citalopram | Placebo
Started | 17 | 16
Completed | 16 | 15
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Citalopram | Placebo | Total
Number analyzed (Participants) | 17 | 16 | 33
Age Continuous [Mean (Standard Deviation); unit: years]
  Age | 47.33 (14.61) | 45.13 (13.59) | 46.2 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Executive Function Composite Score Comparing Visit 2 (Week 0) to Visits 5 (Week 12) & 6 (Week 15) for the Citalopram Cohort Versus Placebo Cohort.
Description: Full Scale Name: The Executive Composite Score (ECS). Definition: Subscales were averaged to compute this composite total score. The ECS is the weighted average of performance on 6 subtests of executive function, including (1) the Controlled Oral Word Association Test, (2) Symbol Digit Modalities test; (3) Stroop Color Word Test (Interference Trial), (4) Trail Making test (Part B), (5) Letter-Number Sequencing, and (6) Animal Naming. Construct Measured: Thinking tasks involving planning, working memory, attention, problem solving, verbal reasoning, inhibition, mental flexibility, and task switching. ECS Scale Range: The ECS score ranges from -5 to +5 on a standardized (Z) score scale, where lower scores indicate poorer performance on executive functioning tasks. Change Calculation Details: Compares change in executive functioning performance from visit 2 (week 0) to the weighted average of visits 5 (week 12) & 6 (week 15) for the citalopram versus placebo cohort.
Time Frame: after 15 weeks of treatment
Population: Intention to treat analysis was performed using a mixed linear model controlling for practice effects comparing visit 2 (week 0) to the weighted average of visits 5 (week 12) & 6 (week 15) for the citalopram versus placebo cohort
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 16 | 15
units on a scale | 0.005 (0.067) | 0.172 (0.071)
Statistical Analysis 1: Comparison: Citalopram vs Placebo; Mixed linear model with treatment-group-specific random subject effects: Predefined 2-tailed linear treatment contrast of intention-to-treat, with Kenward-Rogers correction (t statistic); Test type: Superiority or Other; p = 0.092, 2-tailed linear treatment contrast; This was a predefined 2-tailed linear treatment contrast of intention-to-treat, with Kenward-Rogers correction (t statistic); Mean Difference (Net) = -0.166, 95% CI 2-sided [-0.361 to 0.028], Standard Error of Mean 0.098

2. Secondary Outcome: Letter Number Sequencing Score Comparing Visit 2 (Week 0) to Visits 5 (Week 12) & 6 (Week 15) for the Citalopram Cohort Versus Placebo Cohort
Description: Full Scale Name: Letter Number Sequencing (LNS) subtest from the Wechsler Adult Intelligence Scale (WAIS) third edition. Definition: LNS is a task that requires the reordering of an initially unordered set of letters and numbers. Construct Measured: Working memory. LNS Score Range: Raw scores may range from 0 to 21, where lower scores indicate poorer performance in working memory. Change Calculation Details: Compares change in working memory performance from visit 2 (week 0) to the weighted average of visits 5 (week 12) & 6 (week 15) for the citalopram versus placebo cohort.
Time Frame: after 15 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 16 | 15
units on a scale | -0.113 (0.113) | 0.225 (0.124)
Statistical Analysis 1: Comparison: Citalopram vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.048, 2-tailed linear treatment contrast; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.337, 95% CI 2-sided [-0.672 to -0.003], Standard Error of Mean 0.168

3. Secondary Outcome: Semantic Fluency Score Comparing Visit 2 (Week 0) to Visits 5 (Week 12) & 6 (Week 15) for the Citalopram Cohort Versus Placebo Cohort
Description: Semantic Fluency Score. Definition: The Semantic Fluency Score is the number of words a person can produce given a category, including naming (1) Animal names, (2) Fruit names, (3) Boy names, (4) Girl names, and (5) Vegetable names. Construct Measured: Working memory and verbal initiation. Scale Range: The Semantic Fluency Score ranges from -5 to +5 on a standardized (Z) score scale, where lower scores indicate poorer performance on working memory tasks. Change Calculation Details: Compares change in working memory performance from visit 2 (week 0) where patients named fruit names to the weighted average of visits 5 (week 12) & 6 (week 15) where patients named girl names and vegetable names respectively for the citalopram versus placebo cohort.
Time Frame: after 15 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 16 | 15
units on a scale | 0.386 (0.192) | 0.664 (0.187)
Statistical Analysis 1: Comparison: Citalopram vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.302, 2-tailed linear treatment contrast; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.278, 95% CI 2-sided [-0.810 to 0.254], Standard Error of Mean 0.268

4. Secondary Outcome: Symbol-Digit Modalities Score Comparing Visit 2 (Week 0) to Visits 5 (Week 12) & 6 (Week 15) for the Citalopram Cohort Versus Placebo Cohort
Description: Full Scale Name: The Symbol Digit Modalities Test (SDMT). Definition: The SDMT screens for organic cerebral dysfunction by having the examinee use a reference key to pair specific numbers with given geometric figures in 90 seconds. Construct Measured: Attention, processing speed, and working memory. SDMT Scale Range: Raw scores may range from 0 to 110, where lower scores indicate poorer performance. Change Calculation Details: Compares change in performance from visit 2 (week 0) to the weighted average of visits 5 (week 12) & 6 (week 15) for the citalopram versus placebo cohort.
Time Frame: after 15 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 16 | 15
units on a scale | -0.227 (0.113) | -0.170 (0.103)
Statistical Analysis 1: Comparison: Citalopram vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.708, 2-tailed linear treatment contrast; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.057, 95% CI 2-sided [-0.361 to 0.246], Standard Error of Mean 0.153

5. Secondary Outcome: Verbal Fluency Score Comparing Visit 2 (Week 0) to Visits 5 (Week 12) & 6 (Week 15) for the Citalopram Cohort Versus Placebo Cohort
Description: Full Scale Name: The Verbal Fluency Score (VFC). Definition: The VFC is the number of words a person can produce given a letter, including (1) Naming words that start with F, A, and S; (2) naming words that start with K, W, and R; (3) naming words that start with V, I, and P; (4) naming words that start with O, G, and B; (5) naming words that start with E, N, and T; and (6) naming words that start with J, C, and S. Construct Measured: Verbal initiation and flexibility. Scale Range: The Verbal Fluency Composite Score ranges from -5 to +5 on a standardized (Z) score scale, where lower scores indicate poorer performance. Change Calculation Details: Compares change in verbal initiation and flexibility from visit 2 (week 0) where patients named words starting with O, G, and B to the weighted average of visits 5 (week 12) and 6 (week 15) where patients named words starting with E, N, and T, and J, C, and S respectively for the citalopram versus placebo cohort.
Time Frame: after 15 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 16 | 15
units on a scale | 0.140 (0.109) | 0.071 (0.103)
Statistical Analysis 1: Comparison: Citalopram vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.646, 2-tailed linear treatment contrast; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.069, 95% CI 2-sided [-0.229 to 0.367], Standard Error of Mean 0.150

6. Secondary Outcome: Stroop Interference Score Comparing Visit 2 (Week 0) to Visits 5 (Week 12) & 6 (Week 15) for the Citalopram Cohort Versus Placebo Cohort
Description: Full Scale Name: Stroop Interference subtest from The Stroop Color and Word Test. Definition: Participants are asked to name the ink color in which a word is printed when the word itself (which is irrelevant to the task) is the name of a different color rather than the same color. For example, participants may be asked to say "red" to the word blue printed in red ink. Constructs Measured: Selective attention, response inhibition, cognitive flexibility, and processing speed. Scale Range: The Stroop Interference score ranges from -5 to +5 on a standardized (Z) score scale, where lower scores indicate poorer performance. Change Calculation Details: Compares change in attention and processing speed performance from visit 2 (week 0) to the weighted average of visits 5 (week 12) and 6 (week 15) for the citalopram versus placebo cohort.
Time Frame: after 15 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 16 | 15
units on a scale | -0.256 (0.122) | -0.046 (0.123)
Statistical Analysis 1: Comparison: Citalopram vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.230, 2-tailed linear treatment contrast; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.210, 95% CI [-0.554 to 0.135], Standard Error of Mean 0.174

7. Secondary Outcome: Trails B Score Comparing Visit 2 (Week 0) to Visits 5 (Week 12) & 6 (Week 15) for the Citalopram Cohort Versus Placebo Cohort
Description: Full Scale Name: Trail Making Test Part B (TMT-B). Definition: The TMT-B test requires participants to "connect-the-dots" of 25 consecutive targets on a sheet of paper where the subject alternates between numbers and letters, going in both numerical and alphabetical order. Constructs Measured: Attention, set shifting, and processing speed. Scale range: The TMT-B score ranges from -5 to +5 on a standardized (Z) score scale, where lower scores indicate poorer performance. Change Calculation Details: Compares change in attention and processing speed performance from visit 2 (week 0) to the weighted average of visits 5 (week 12) and 6 (week 15) for the citalopram versus placebo cohort.
Time Frame: after 15 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 16 | 15
units on a scale | 0.087 (0.273) | 0.405 (0.397)
Statistical Analysis 1: Comparison: Citalopram vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.512, 2-tailed linear treatment contrast; [statistical method as in outcome 1, analysis 1]; Median Difference (Net) = -0.317, 95% CI 2-sided [-1.276 to 0.642], Standard Error of Mean 0.482

8. Secondary Outcome: Hamilton Rating Scale for Depression Comparing Screening (Intake Visit) to Visit 6 (Week 15) for the Citalopram Cohort Versus Placebo Cohort
Description: Full Scale Name: Hamilton Rating Scale for Depression (HAM-D). Definition: The Hamilton Rating Scale for Depression is a clinician-administered multiple item questionnaire used to provide an indication of depression. Construct Measured: Depression. HAM-D Score Range: Raw scores may range from 0 to 54, where higher scores indicate worsening mood. Change Calculation Details: Compares change in mood from screening (intake visit) to visit 6 (week 15) for the citalopram versus placebo cohort.
Time Frame: after 15 weeks of treatment
Population: Intention to treat analysis was performed using a mixed linear model comparing screening (intake visit) to Visit 6 (week 15) for the citalopram versus placebo cohort
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 16 | 15
units on a scale | -0.67 (0.76) | 1.23 (0.89)
Statistical Analysis 1: Comparison: Citalopram vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.12, 2-tailed linear treatment contrast; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -1.90, 95% CI 2-sided [-4.30 to 0.50], Standard Error of Mean 1.17

9. Secondary Outcome: Total Functional Capacity Score Comparing Baseline (Week -4) to Visits 4 (Week 6) & 6 (Week 15) for the Citalopram Cohort Versus Placebo Cohort
Description: Full Scale Name: The Total Functional Capacity (TFC) subscale from the Unified Huntington's Disease Rating Scale (UHDRS). Definition: The TFC is a score that classifies five stages of Huntington's Disease and five levels of function in the domains of workplace, finances, domestic chores, activities of daily living and requirements for unskilled or skilled care. Construct Measured: Activities of Daily Living. Scale Range: The TFC score ranges from 0 to 13, where lower scores indicate poorer performance in activities of daily living. Change Calculation Details: Compares change in TFC performance from Baseline (week -4) to the weighted average of visits 4 (week 6) and 6 (week 15) for the citalopram versus placebo cohort.
Time Frame: after 15 weeks of treatment
Population: Intention to treat analysis was performed using a mixed linear model comparing baseline (week -4) to the weighted average of Visits 4 (week 6) & 6 (week 15) for the citalopram versus placebo cohort
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 16 | 15
units on a scale | -0.54 (0.46) | -0.06 (0.50)
Statistical Analysis 1: Comparison: Citalopram vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.49, 2-tailed linear treatment contrast; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.48, 95% CI 2-sided [-1.87 to 0.91], Standard Error of Mean 0.68

10. Secondary Outcome: Subgroup Analysis of the Hamilton Depression Rating Scale Comparing Screening (Intake Visit) to Visit 6 (Week 15) for the Citalopram Cohort Versus Placebo Cohort
Description: Full Scale Name: Hamilton Rating Scale for Depression (HAM-D). Definition: The Hamilton Rating Scale for Depression is a clinician-administered multiple item questionnaire used to provide an indication of depression. Construct Measured: Depression. HAM-D Score Range: Raw scores may range from 0 to 54, where higher scores indicate worsening mood. Change Calculation Details: This analysis was restricted to a subgroup and, accordingly, does not reflect the total number of participants as reported in the Participant Flow. This analysis compares change in mood from screening (intake visit) to visit 6 (week 15) for the citalopram versus placebo cohort.
Time Frame: after 15 weeks of treatment
Population: This analysis was restricted to a subgroup and, accordingly, does not reflect the total number of participants as reported in the Participant Flow. This analysis compares change in mood from screening (intake visit) to visit 6 (week 15) for the citalopram versus placebo cohort.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 14 | 14
units on a scale | -0.10 (0.85) | 1.50 (0.9)
Statistical Analysis 1: Comparison: Citalopram vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis — Predefined 2-tailed linear treatment contrast of intention-to-treat, with Kenward-Rogers correction (t statistic); Odds Ratio (OR) = -2.5, 95% CI 2-sided [-5.04 to 0.04], Standard Error of Mean 1.23

ADVERSE EVENTS:
Time Frame: A systematic assessment of adverse experiences was captured at every encounter beginning at Visit 2 (week 0) and continuing through Visit 7 (week 16) for the randomized treatment vs. placebo period.
Description: 17 Participants were randomized to citalopram and 16 participants were randomized to placebo, using a 1:1 allocation.
Arm/Group | Citalopram | Placebo
Serious Adverse Events (participants affected / at risk) | 1/17 | 2/16
Other Adverse Events (participants affected / at risk) | 6/17 | 3/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Citalopram (N=17) | Placebo (N=16)
worsening depression with suicidal ideation (Psychiatric disorders) | 1 (1) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Citalopram (N=17) | Placebo (N=16)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Ejaculation Disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Insomnia (General disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Statistical power was limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No